CLINICAL TRIAL: NCT00772772
Title: The Effect of Vitamin D3 Repletion in Chronic Kidney Disease Stage 3
Brief Title: Vitamin D Repletion in Chronic Kidney Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Manish Ponda, Assistant Professor of Clinical Investigation, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAP-0626
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Kidney Disease
Keywords: Vitamin D3 repletion; levels of endotoxin; intestinal permeability; accelerated atherosclerosis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3 (Experimental): Vitamin D3 30,000 international units orally per week for 8 weeks
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — 2 single oral dose of Vitamin D3 30,000 international units and 8 weeks supply of Vitamin D3 (10,000 IU tablets, 3 pills to be taken by mouth as one dose weekly)
  Other Names: Vitamin D

SUMMARY:
The reason for doing this research is that people with kidney disease often suffer from heart disease. Why this happens is not fully known. A possible cause may be high blood levels of a substance made by bacteria called "endotoxin". The blood levels of this substance are high in people with medium-level kidney disease.

We want to know if replacing normal amounts of Vitamin D can help lower the levels of this substance. We also want to know if replacing normal amounts of Vitamin D is associated with other changes that may help heart disease. We hope that our research will help figure out if levels of this substance can be lowered by replacing normal amounts of Vitamin D. Normal subjects are enrolled to have a 'control' set for comparison purposes.

DETAILED DESCRIPTION:
Your participation in this study requires:

* 4 visits to the outpatient clinic (including 1 screening visit)
* Providing a blood sample (less than 5 tablespoons) and a urine sample at each visit
* Taking a test to measure how leaky your gut is. This test requires that you drink a small amount of liquid (about 4 ounces) and then collect your urine for 6 hours after drinking the liquid.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy volunteers

* Males and post-menopausal females, between the age of 50 -80.
* Vitamin D 25-OH level less than 20 ng/ml

Inclusion Criteria for Medium-level Kidney Function volunteers

* Males and post-menopausal females, between the age of 50 -80.
* Chronic kidney disease stage 3
* Vitamin D 25-OH level less than 20 ng/ml

Exclusion Criteria:

* Serum calcium level >10.5 mg/dl
* Serum phosphorus level > 5.5 mg/dl
* Serum PTH level < 35 pg/ml
* Active infection including HIV, Hepatitis B or C
* History of recent acute infection ( within 1 month)
* Gastrointestinal disease resulting in significant GI dysfunction or malabsorption
* Hgb< 10 g/dL
* Current use of Coumadin
* Current use of Vitamin D >400 IU/day
* Current use of systemic steroids or other immunosuppressants
* History of malignancy not in remission (>6 months)
* History of current ethanol abuse or illicit drug use
* History of significant emotional disorder within the past 5 years
* Participation in an investigational drug study within one month of screening
* Have any other condition, which in the opinion of the investigator, should prohibit the participation in the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Ponda, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3: Vitamin D3 30,000 units PO weekly for 8 weeks
Period: Overall Study
Arm/Group | Vitamin D3
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D3
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Endotoxin Activity
Description: Endotoxin Activity as measured by the Endotoxin Activity Assay. This measurement was made at baseline and after 8 weeks of therapy with Vitamin D3. The measurement of the assay is unitless. It is not based on an absolute amount of endotoxin, but rather the proportion of the theoretical maximal response of the patient and ranges from 0 (lowest) to 1 (highest).
Time Frame: baseline and 8 weeks
Population: Per protocol. Result is expressed as change in endotoxin activity with therapy
Measure: Mean (Standard Deviation); unit: EA units
Groups:
- Patients With Chronic Kidney Disease (CKD): CKD patients who were Vitamin D deficient and received Vitamin D3 repletion
Arm/Group | Patients With Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 12
EA units | -.057 (.018)

2. Secondary Outcome: Blood Pressure
Time Frame: after 8 weeks of vitamin D therapy
Reporting Status: Not Posted

3. Secondary Outcome: Intestinal Permeability
Time Frame: after 8 weeks of vitamin D therapy
Reporting Status: Not Posted

4. Secondary Outcome: Nuclear Magnetic Resonance (NMR) Lipoprotein Profile
Time Frame: after 8 weeks of vitamin D therapy
Reporting Status: Not Posted

5. Secondary Outcome: 25-hydroxy Vitamin D (25-OH Vitamin D)
Description: 25-OH Vitamin D levels were measured in patients with chronic kidney disease at baseline and after 8 weeks of treatment with Vitamin D3 30000 units weekly.
Time Frame: after 8 weeks of vitamin D therapy
Population: Patients with chronic kidney disease had 25-OH vitamin D levels measured at baseline and after 8 weeks of Vitamin D3 therapy. Analysis was per protocol.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | CKD Patients
Number analyzed (Participants) | 12
ng/ml | 37.4 (3.0)

6. Secondary Outcome: 1, 25-OH Vitamin D
Time Frame: after 8 weeks of vitamin D therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Vitamin D3 (N=12)
Metabolic (Metabolism and nutrition disorders) | 2/2 (2)
Cardiovascular (Cardiac disorders) | 1/1 (1)
Hematologic (Blood and lymphatic system disorders) | 1/1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes